CLINICAL TRIAL: NCT02556424
Title: Efficacy and Tolerance Comparison Between Subconjunctival Injection of Triamcinolone and Intravitreal Implant of Dexamethasone for the Treatment of Inflammatory Macular Edema
Acronym: TRIOZ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0056
Record Dates: First submitted 2015-05-29; First posted 2015-09-22 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2020-10

CONDITIONS: Inflammatory Macular Edema
Keywords: Ophthalmology; Uveitic macular edema; Triamcinolone subconjunctival injection; Dexamethasone intraocular implant
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reference Drug (Active Comparator): Intravitreal implant of 700μg of dexamethasone (Ozurdex®)
  Interventions: Drug: Dexamethasone
- Tested Drug (Experimental): Subconjunctival injection of 16 mg triamcinolone (Kénacort Retard®)
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Dexamethasone — Intravitreal implant at D0
  Other Names: Ozurdex®
  Arms: Reference Drug
Drug: Triamcinolone — Subconjunctival injection at 4 mm from the limbus at 6 o'clock
  Other Names: Kénacort retard®
  Arms: Tested Drug

SUMMARY:
Corticosteroids, whether injected peri- or intra-ocularly, remain indispensable tools of the therapeutic arsenal in treating inflammatory macular edema. However, a few years ago, only triamcinolone acetonide was available to ophthalmologists. This molecule, developed initially for rheumatological or dermatological use, has been increasingly deployed in ophthalmology, while still off-label.

In 2011, the delivery system of dexamethasone from biodegradable and injectable implant into the vitreous cavity obtained the label for inflammatory macular edema. This protocol is therefore designed to compare the efficacy and safety of peri- and intra-ocular injections of corticosteroids in the treatment of inflammatory macular edema.

DETAILED DESCRIPTION:
This research compares the implantation techniques of corticosteroids in the eye, with two groups of equal size being followed. This is a multi-center, controlled study, with the reference drug being the intravitreal implant of 700μg of dexamethasone (Ozurdex®) compared to subconjunctival injection of triamcinolone (Kénacort retard®). This is an open, prospective, randomized study. It is not possible, for technical reasons, to inject blind two products with different injection routes and that are visible to the investigator during control examinations (sub-conjunctival crystals and intravitreal implant). However, the assessment of visual acuity and central macular thickness will be performed by an uninformed ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female (under effective contraception if premenopausal) over 18 years old
* Patient affiliated with a social security plan
* Patient able to understand and follow the instructions of the study
* Patient having signed an informed consent
* Patient having a central macular thickness greater than 320μm (Spectral Domain, 270µm Time Domain)
* Patient with an inflammatory macular edema, unilateral or bilateral (in the case of a bilateral inflammatory macular edema, the eye most affected will be treated)

Exclusion Criteria:

* Patient with an infectious uveitis
* Patient with uncontrolled active infection
* Patient receiving an unbalanced general anti-inflammatory and/or immunosuppressive and/or immunomodulatory therapy (recent modification <1 month)
* Patient having a history of glaucoma and/or ocular hypertension in the eye studied (intraocular pressure (IOP) > 25 mmHg without antiglaucoma medication or > 21 mmHg with antiglaucoma combination therapy) and/or cortisone-causing-hypertension not controlled by an antiglaucoma dual therapy
* Patient with uncontrolled diabetes (HbA1c> 8%) or unbalanced hypertension (Systolic Blood Pressure > 160 mmHg and/or Diastolic Blood Pressure > 100mmHg)
* Edematous diabetic maculopathy
* Patient who had received triamcinolone (subconjunctivally or sub-tenon) 3 months before randomization, or 700μg dexamethasone intravitreally 6 months before randomization
* Suspected or active ocular or periocular infection, including most viral diseases of the cornea and conjunctiva, such as active epithelial keratitis with herpes simplex (dendritic keratitis), vaccinia, varicella, mycobacterial infections and mycoses
* History of ocular herpes infection or central serous chorioretinopathy
* Aphakic eye with rupture of the posterior lens capsule
* Eye with implant in the anterior chamber, iris- or transscleral-fixated intraocular implant and rupture of the posterior lens capsule
* Uncontrolled systemic inflammatory disease.
* Known hypersensitivity to the active substance or to one of the excipients of Ozurdex®, Kenacort® or injectable fluorescein
* Pregnant woman or likely to become pregnant or nursing
* Patient participating in another clinical trial
* Adult under a legal protection regime (guardianship, trusteeship, "sauvegarde de justice")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of a subconjunctival injection of triamcinolone on reducing the central macular thickness versus an intravitreal implant of dexamethasone between patient selection and 2 months after treatment | At 2 months after treatment
  Difference of the central macular thickness in the treated eye, measured by Optical Coherence Tomography (OCT) spectral domain, for each patient between patient selection and 2 months after treatment

SECONDARY OUTCOMES:
Evaluation of the experience of the injection by a questionnaire (tolerable, unpleasant and very unpleasant) and by EVA (0 cm = no pain to 10 cm = extreme pain) | At day 0 (= the day of the treatment)
  Scale of "patient experience" the day of the injection (tolerable, unpleasant, very unpleasant) and visual analogue scale (VAS)
Evaluation of the effectiveness of the studied injection at each visit regarding gain in visual acuity (ETDRS) | Up to 6 months
  Visual acuity (ETDRS)
Evaluation of the effectiveness of the studied injection at each visit regarding reduction of the anterior flare | Up to 6 months
  Anterior flare ("Lampe A Fente" and Laser Flare Meter, if available)
Evaluation of the effectiveness of the studied injection at each visit regarding reduction of the vitreous haze | Up to 6 months
  Vitreous flare
Evaluation of the effectiveness of the studied injection at each visit regarding central macular thickness measured by OCT, allowing the evaluation of the duration of action of the treatment | Up to 6 months
  Central macular thickness of the eye treated for determining the duration of action
Evaluation of the effectiveness of the studied injection at each visit regarding local and general tolerance, by collecting all Adverse Events (AEs) / Serious Adverse Events (SAEs) | Up to 6 months
  Evaluation of tolerance by collecting all AEs / SAEs of randomized patients, such as intra-ocular hypertension, cataracts, endophthalmitis, poor glycemic and/or blood pressure control
Evaluation of the effectiveness of the studied injection at each visit regarding patients' quality of life | Up to 6 months
  Patients' quality of life questionnaire (EQ-5D)

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - CHU Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Dijon, Dijon
  - CHU de Grenoble, La Tronche
  - Hôpital Bicêtre (AP-HP), Le Kremlin-Bicêtre
  - CHRU de Lille, Lille
  - Hopices Civils de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - Hôpital La Pitié-Salpêtrière (AP-HP), Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
  - CHU de Tours, Tours
  - CHU de Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Couret C, Poinas A, Volteau C, Riche VP, Le Lez ML, Errera MH, Creuzot-Garcher C, Baillif S, Kodjikian L, Ivan C, Le Jumeau de Kergaradec LM, Chiffoleau A, Jobert A, Jaulin J, Biron L, Hervouet E, Weber M. Comparison of two techniques used in routine care for the treatment of inflammatory macular oedema, subconjunctival triamcinolone injection and intravitreal dexamethasone implant: medical and economic importance of this randomized controlled trial. Trials. 2020 Feb 10;21(1):159. doi: 10.1186/s13063-020-4066-0. PMID 32041669